CLINICAL TRIAL: NCT05530512
Title: Neuroimmune Mechanisms Underlying Electroacupuncture Effect on Vascular Function
Brief Title: Acupuncture Therapy and Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Shaista Malik, Professor, University of California, Irvine
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: 19992222; R01AT011306 (NIH)
Record Dates: First submitted 2022-08-27; First posted 2022-09-07 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Mild to Moderate Hypertension
Keywords: hypertension, electroacupuncture
MeSH Terms: conditions — Hypertension | interventions — Electroacupuncture; Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: two by two factorial design for a 4 arm study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The pharmacologist who assays the plasma and serum is masked in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Anti-inflammatory EA (AI-EA) (Experimental): Anti-inflammatory electroacupuncture therapy
  Interventions: Other: electroacupuncture
- Sympathoinhibitory EA (SI-EA) (Experimental): sympatho-inhibitory electroacupuncture therapy
  Interventions: Other: electroacupuncture
- Combined EA (cEA) (Experimental): combination of SI-EA and AI-EA
  Interventions: Other: electroacupuncture
- Control EA (Sham-EA) (Experimental): Sham electroacupuncture
  Interventions: Other: electroacupuncture

INTERVENTIONS:
Other: electroacupuncture — acupuncture needling and stimulation are applied for 30 min
  Other Names: acupuncture

SUMMARY:
Acupuncture therapy will be provided to reduce blood pressure in hypertensive patients. The mild to moderate hypertensive patients will be either on or off hypertensive medications. The course last for 8 weeks and the frequency is once a week.

DETAILED DESCRIPTION:
Improvement in BP control rates would lead to one of the largest impacts in improving life expectancy and the quality of life for over 100 million people in the United States and 1 billion people worldwide with immediate and measurable results. In the United States, 80% of patients with HTN are treated, but BP is controlled in only half of these individuals, with control worsening with increasing age. The reasons for inadequate treatment and BP control are complex, but one reason for this therapeutic misalignment may be an incomplete understanding of the mechanisms underlying the development and progression of HTN. The aging process leads to dysfunction of the ANS, resulting in neuroendocrine abnormalities and chronic low-grade inflammation.

The investigators have previously shown that electroacupuncture (EA) at four targeted acupoints, can decrease sympathetic activity [sympathoinhibitory (SI)], approaching levels close to those present prior to onset of HTN and may address this unmet need in HTN management. The investigators are now testing and have preliminary evidence that EA at two additional acupoints (SP6-7) increases parasympathetic activation, thereby decreasing circulating and tissue inflammatory biomarkers [thus anti-inflammatory (AI)] and when combined with SI-EA can improve measures of vascular health including endothelial function and arterial stiffness in preclinical model with overall greater reduction in BP. Together these combined six acupoints, when simultaneously activated by EA may restore optimal autonomic control of the immune system and target an important mechanistic pathway not addressed by BP-lowering pharmacotherapy alone. To date, 39 participants have been enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects from 45 to 75 years of age
2. Clinically diagnosed with mild to moderate hypertension and ON or OFF medication (Office SBP > 140 mmHg and < 160 mmHg Or ABPM average SBP > 130 mmHg and < 145 mmHg), and
3. No significant ECG change reflecting ischemia (i.e. ST elevation or depression) at rest will be recruited to participate in this study.

Exclusion Criteria:

1. Subjects will be excluded if pregnant or nursing.
2. Subjects will be excluded if they have coronary disease (by history or on ECG screening), conduction abnormalities on ECG consistent with left bundle branch block, cardiac arrhythmias associated with low blood pressure (<90 mmHg), peripheral vascular disease, orthopedic disease, diabetic neuropathy or severe hypertension (BP >170 mmHg systolic or >110 mmHg diastolic), or any other physical or psychological illness.
3. Those with known sensitivity to any topical preparations or strong reactions to medical dressings and skin tapes also will be excluded.
4. Inability our or unwillingness of individual to give written informed consent.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in sympathetic and parasympathetic nervous systems | through study completion, an average of 4.5 years
  Heart rate variability and its component will be evaluated with EKG.

SECONDARY OUTCOMES:
Change in biomarkers like cytokines | through study completion, an average of 4.5 years
  Plasma will be measured for inflammatory markers with ELISA kits.

OTHER OUTCOMES:
Change in blood pressure | through study completion, an average of 4.5 years
  Blood pressure (systolic and diastolic) will be measured with an ambulatory blood pressure device every 20 min for 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Shaista Malik, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - Susan Samueli Integrative Health Institute, Irvine, California
  - University of California, Irvine, Health Sciences Medical Center, Orange, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: animal study — https://doi.org/10.3389/fcvm.2023.1140255